CLINICAL TRIAL: NCT06665438
Title: Impact of Dexmedetomidine Add to Intra-articular Bupivacaine for Post Operative Analgesia After Knee Arthroscopic Surgery
Brief Title: Dexmedetomidine and Bupivacaine Intra-articular for Postoperative Analgesia After Knee Arthroscopic Surgery
Acronym: DEXMED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Mahmoud, Lecturer of anesthesia, intensive care and pain management, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZAST/Research/88/14-MAY-2024.
Record Dates: First submitted 2024-10-21; First posted 2024-10-30 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Analgesia
Keywords: Knee arthroscopy; Bupivacaine; Dexmedetomidine; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: patients randomly allocate to one of three groups (n =25) for intra articular injection using Sealed envelope method as follows: Group (C), receive 18 ml saline only and serve as the control group(C). Group (B) receive 18ml 0.25% bupivacaine. Group(D)received 18 ml 0.25% bupivacaine and dexmedetomidine 1 μg/kg, the study drugs will injected in the knee joint by the surgeon through the arthroscope after completing the procedure (without knowing the drugs used)
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group of control (C) (Experimental): receive 18 ml of normal saline only and serve as the control group.the normal saline will injected in the knee joint by the surgeon through the arthroscope after completing the procedure
  Interventions: Drug: Normal Saline (Placebo)
- groups of Bupivacaine (B) (Experimental): The 18ml 0.25% bupivacaine will injected intra articular in the knee joint by the surgeon through the arthroscope after completing the procedure
  Interventions: Drug: Bupivacaine 0.25%; Drug: Dexmedetomidine
- groups of dexmedetomidine (D) (Experimental): Dexmedetomidine 1 μg/kg will injected intra articular in the knee joint by the surgeon through the arthroscope after completing the procedure.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Normal Saline (Placebo) — the 18 ml of normal saline will injected intra articular in the knee joint by the surgeon through the arthroscope after completing the procedure
  Arms: group of control (C)
Drug: Bupivacaine 0.25% — the 18ml 0.25% bupivacaine. will injected intra articular in the knee joint by the surgeon through the arthroscope after completing the procedure
  Arms: groups of Bupivacaine (B)
Drug: Dexmedetomidine — Dexmedetomidine 1 μg/kg will injected intra articular in the knee joint by the surgeon through the arthroscope after completing the procedure.
  Arms: groups of Bupivacaine (B); groups of dexmedetomidine (D)

SUMMARY:
The aim of this study to compare the analgesic effects of intraarticular dexmedetomidine added to bupivacaine with those of bupivacaine alone after knee arthroscopy

DETAILED DESCRIPTION:
prospective double-blind study perform on 75 patients candidates for anterior cruciate ligament (ACL) reconstruction by knee arthroscopy refer to the clinic of Al Azhar University Hospital, Assiut, Egypt, to evaluate the effect of adding dexmedetomidine to intra articular bupivacaine injection on postoperative pain after knee arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Either sex
* Aged 18-65 years
* Candidates for anterior cruciate ligament (ACL) reconstruction by knee arthroscopy
* Exclusion Criteria:
* the patients with kidney failure, liver failure, valvular and ischemic heart disease , high blood pressure, diabetes, history of infection and malignancy.
* history of coagulation diseases, and history of drug allergies to used drugs.
* those who consumed NSAIDs and analgesics 24 h before surgery were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change on the visual analog scale (VAS) for pain (0 = no pain to 100 = the maximum pain )to assessment the duration of analgesia following the surgery | post operative at 30 minute, 1 hour, 2 hour, 4 hour, 6 hour, 12 hour, and 24 hour .
  Change on the visual analog scale (VAS) for pain (0 = no pain to 100 = the maximum pain) to assessment the duration of analgesia following intra articular injection of Bupivacaine and Dexmedetomidine after knee arthroscopy

SECONDARY OUTCOMES:
Total meperidine consumption . Meperidine will be used intravenously if the visual analog scale ( VAS) score was >50 to control postoperative pain. | The total dose of meperidine given between the study groups during the first 24 hour( post operative at 30 minute, 1 hour, 2 hour, 4 hour, 6 hour, 12 hour, and 24 hour),will be recorded.
  the secondary outcome variables will be the total dose of meperidine given between the study groups.Meperidine will be used intravenously if the visual analog scale ( VAS) score was >50 to control postoperative pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No